CLINICAL TRIAL: NCT00843193
Title: A Multi-Centre, Randomized, Double-Blind, Placebo-Controlled, Repeat-Dose Study to Evaluate the Efficacy and Safety of Intravenous GSK679586 in Patients With Severe Asthma
Brief Title: Efficacy and Safety Study of GSK679586 in Patients With Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 106870
Record Dates: First submitted 2009-02-05; First posted 2009-02-13 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Asthma
Keywords: Asthma; Asthma control questionnaire
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK679586 (Experimental): Subjects will receive three, once monthly intravenous administration of 10 mg/kg of GSK679586, according to randomization
  Interventions: Drug: INTRAVENOUS GSK679586; Drug: FLUTICASONE PROPIONATE
- PLACEBO (Placebo Comparator): Subjects will receive three, once monthly intravenous administration of saline, according to randomization
  Interventions: Drug: INTRAVENOUS PLACEBO; Drug: FLUTICASONE PROPIONATE

INTERVENTIONS:
Drug: INTRAVENOUS GSK679586 — GSK679586 will be provided as a clear or colorless to pale yellow liquid with the unit dose strength of 10mg/kg and will be infused over an hour. The infusion will be delivered by a programmable infusion pump
  Arms: GSK679586
Drug: INTRAVENOUS PLACEBO — Clear or colorless 0.9% sodium chloride saline solution will be infused over an hour. The infusion will be delivered by a programmable infusion pump
  Arms: PLACEBO
Drug: FLUTICASONE PROPIONATE — Subjects will be supplied fluticasone propionate at Screening, Run-in and when needed during the study. Subjects will be up-titrated to 1000 μg/day and those who were already taking greater than equal to 1000 μg/day fluticasone propionate or equivalent prior to the study will remain on their pre-study dose.

SUMMARY:
Treatment, Randomised, Double Blind, Parallel Assignment, Safety/efficacy Study

DETAILED DESCRIPTION:
A Multi-Centre, Multi-country, Randomized, Double-Blind (Subject, Investigator), Placebo-Controlled, Repeat-Dose study to evaluate the Efficacy and Safety of Intravenous GSK679586 in Patients with Severe Asthma

ELIGIBILITY:
Inclusion Criteria:

* history of asthma for ≥ 6 months
* taking inhaled corticosteroids
* non-smoking
* Baseline (pre-bronchodilator) FEV1 35-80% predicted at screening.
* Reversible airways disease as indicated by an increase of FEV1 ≥12% from baseline after nebulised salbutamol or albuterol.
* symptomatic according to the ACQ-7

Exclusion Criteria:

* Unstable severe asthma
* Recent respiratory illness
* Presence of other respiratory disease or chronic pulmonary condition other than asthma
* Treatment with omalizumab within 4 months of study
* Recent gastrointestinal or respiratory parasitic infestation
* History of severe allergy to food or drugs

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2008-12-09 (Actual); Primary Completion 2010-07-25 (Actual); Study Completion 2010-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- United States (6):
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Madison, Wisconsin
- France (7):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Saint-Pierre
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Tarbes
- Germany (3):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
- Netherlands (3):
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hoorn
- Norway (2):
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Trondheim
- Poland (5):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Gidle
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Warsaw
- South Africa (4):
  - GSK Investigational Site, Cape Town, Gauteng
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Mowbray
- United Kingdom (5):
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, Guildford, Surrey
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Anderson WH, Koshy BT, Huang L, Mosteller M, Stinnett SW, Condreay LD, Ortega H. Genetic analysis of asthma exacerbations. Ann Allergy Asthma Immunol. 2013 Jun;110(6):416-422.e2. doi: 10.1016/j.anai.2013.04.002. PMID 23706709
- See also: Ginasthma.com is a website of the Global Initiative for Asthma. This study uses the GINA guidance, 2007 for diagnosis asthma patients who are eligible for entry this study. — http://www.ginasthma.com/
- Available data/document: Study Protocol: 106870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in participants with severe asthmatics from 9-Dec-2008 to 19-July-2010 at 35 study centers in France (7), United States (6), United Kingdom (5), Poland (5), South Africa (4), Germany (3), Netherlands (3) and Norway (2).
Pre-assignment Details: During run-in period of 28 days each participant's inhaled corticosteroid (ICS) dose was up-titrated to 1000 microgram (μg)/day fluticasone propionate. Participants already taking ≥ 1000 µg/day fluticasone propionate or equivalent prior to study remained on their pre-study dose. Total of 198 participants were randomized and treated in the study.
Groups:
- Placebo: Participants received a total of three once-monthly intravenous (IV) infusions of sodium chloride placebo in a volume matched to the volume that would had been administered if the participant had been randomized to active treatment in order to maintain the integrity of the study blind. The IV infusions were administered by qualified study personnel, and were administered over 1 hour using a programmable infusion pump.
- GSK679586 10mg (Milligram)/kg(Kilogram): Participants received a total of 3 once-monthly IV infusions of 10 mg/kg GSK679586 diluted with sterile, normal saline to a concentration of 25 mg/ milliliter (mL). The final solution volume was 40 to 60 mL, depending on participants weight. The IV infusions were administered by qualified study personnel, and were administered over 1 hour using a programmable infusion pump.
Period: Overall Study
Arm/Group | Placebo | GSK679586 10mg (Milligram)/kg(Kilogram)
Started | 99 | 99
Completed | 91 | 88
Not Completed | 8 | 11
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received a total of three once-monthly IV infusions of sodium chloride placebo in a volume matched to the volume that would had been administered if the participant had been randomized to active treatment in order to maintain the integrity of the study blind. The IV infusions were administered by qualified study personnel, and were administered over 1 hour using a programmable infusion pump.
- GSK679586 10 mg/kg: Participants received a total of 3 once-monthly IV infusions of 10 mg/kg GSK679586 diluted with sterile, normal saline to a concentration of 25 mg/mL. The final solution volume was 40 to 60 mL, depending on participants weight. The IV infusions were administered by qualified study personnel, and were administered over 1 hour using a programmable infusion pump.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK679586 10 mg/kg | Total
Number analyzed (Participants) | 99 | 99 | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.2 (11.78) | 51.2 (11.13) | 51.2 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 51 | 100
  Male | 50 | 48 | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 3 | 1 | 4
  Japanese/East Asian/South East Asian | 0 | 2 | 2
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White | 95 | 96 | 191

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-7) Over 12 Weeks
Description: The ACQ-7 consists of 7 questions scored between zero (no impairment/ limitation) to 6 (total impairment/ limitation). The values of Week 1 is considered as Baseline. ACQ-7 was calculated as the average of the 7 scores. If any one individual score was missing, the ACQ-7 was set to missing.The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well.
Time Frame: Baseline to Week 12
Population: Intent-to-Treat (ITT) population was comprised of all participants who are randomized and receive at least the first dose of study medication. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on Scale
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Scores on Scale
  Week 2: number analyzed (Participants) | 97 | 97
  Week 2 | -0.1 (0.06) | -0.2 (0.06)
  Week 4: number analyzed (Participants) | 95 | 94
  Week 4 | -0.1 (0.06) | -0.3 (0.05)
  Week 8: number analyzed (Participants) | 92 | 92
  Week 8 | -0.2 (0.07) | -0.3 (0.07)
  Week 12: number analyzed (Participants) | 91 | 90
  Week 12 | -0.3 (0.08) | -0.4 (0.09)
Statistical Analysis 1: Comparison: Placebo vs GSK679586 10 mg/kg; Comparison between GSK679586 10 mg/kg and Placebo at Week 2; Test type: Superiority or Other; p = 0.1955, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.27 to 0.06]
Statistical Analysis 2: Comparison: Placebo vs GSK679586 10 mg/kg; Comparison between GSK679586 10 mg/kg and Placebo at Week 4; Test type: Superiority or Other; p = 0.0193, Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.34 to -0.03]
Statistical Analysis 3: Comparison: Placebo vs GSK679586 10 mg/kg; Comparison between GSK679586 10 mg/kg and Placebo at Week 8; Test type: Superiority or Other; p = 0.6156, Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.23 to 0.14]
Statistical Analysis 4: Comparison: Placebo vs GSK679586 10 mg/kg; Comparison between GSK679586 120 mg/kg and Placebo at Week 12; Test type: Superiority or Other; p = 0.4672, ANCOVA; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.31 to 0.14]

2. Secondary Outcome: Change From Baseline in ACQ-7 Over 16 Weeks and 24 Weeks
Description: The ACQ-7 is a 7-item questionnaire that provides a measure of a participant's asthma control. Participant responses were recorded on a 7-point scale ranging from zero (no impairment/ limitation) to 6 (total impairment/ limitation). The values of Week 1 is considered as Baseline. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well. Change from Baseline of Week 16 and Week 24 are incorporated here which are Follow up weeks.
Time Frame: Week 16 and Week 24
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on Scale
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Scores on Scale
  Week 16: number analyzed (Participants) | 92 | 90
  Week 16 | -0.3 (0.08) | -0.4 (0.08)
  Week 24: number analyzed (Participants) | 96 | 95
  Week 24 | -0.3 (0.09) | -0.2 (0.08)

3. Secondary Outcome: Number of Participants Who Demonstrated a Clinically Meaningful Change in ACQ-7 Over the 12 Weeks Assessment Period.
Description: The ACQ-7 is a 7-item questionnaire that provides a measure of a participant's asthma control. Participant responses were recorded on a 7-point scale ranging from zero (no impairment/ limitation) to 6 (total impairment/ limitation). The percentage of participants who were classified as responders for ACQ-7, defined as a clinically meaningful decrease from baseline in ACQ-7 of at least 0.50, was generally similar between treatment groups at each visit and over the 12-week treatment period.
Time Frame: Upto 12 weeks
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Participants
  Week 2: number analyzed (Participants) | 98 | 97
  Week 2 | 16 | 20
  Week 4: number analyzed (Participants) | 96 | 94
  Week 4 | 22 | 29
  Week 8: number analyzed (Participants) | 94 | 92
  Week 8 | 31 | 26
  Week 12: number analyzed (Participants) | 93 | 91
  Week 12 | 33 | 36

4. Secondary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) Over 12 Weeks.
Description: FEV1 is forced expiratory volume in 1 second.Change from Baseline FEV1 was calculated for each of the following visit: Visit 6, Visit 7, Visit 9 and Visit 11. A binary variable was created for each participant with 1 for the responder and 0 for the non nonresponder at each visit. Week 1 was considered as the Baseline. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well.
Time Frame: Baseline to Week 12
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Millilitre (mL)
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Millilitre (mL)
  Week 2: number analyzed (Participants) | 98 | 97
  Week 2 | 0.009 (0.0275) | 0.002 (0.0277)
  Week 4: number analyzed (Participants) | 96 | 93
  Week 4 | 0.033 (0.0331) | 0.037 (0.0288)
  Week 8: number analyzed (Participants) | 93 | 91
  Week 8 | 0.035 (0.0335) | -0.009 (0.0313)
  Week 12: number analyzed (Participants) | 91 | 90
  Week 12 | 0.078 (0.0331) | -0.016 (0.0373)
Statistical Analysis 1: Comparison: Placebo vs GSK679586 10 mg/kg; Comparison between GSK679586 10 mg/kg and Placebo at Week 2; Test type: Superiority or Other; p = 0.7693, ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.08 to 0.06]
Statistical Analysis 2: Comparison: Placebo vs GSK679586 10 mg/kg; Comparison between GSK679586 10 mg/kg and Placebo at Week 4; Test type: Superiority or Other; p = 0.8987, Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.08 to 0.09]
Statistical Analysis 3: Comparison: Placebo vs GSK679586 10 mg/kg; Comparison between GSK679586 10 mg/kg and Placebo at Week 8; Test type: Superiority or Other; p = 0.4231, Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.12 to 0.05]
Statistical Analysis 4: Comparison: Placebo vs GSK679586 10 mg/kg; Comparison between GSK679586 10 mg/kg and Placebo at Week 12; Test type: Superiority or Other; p = 0.0537, Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.19 to 0.00]

5. Secondary Outcome: Change From Baseline in FEV1 Over 16 Weeks and 24 Weeks
Description: FEV1 is forced expiratory volume in 1 second.Change from Baseline FEV1 was calculated for each of the following visit: Visit 6, Visit 7, Visit 9 and Visit 11. A binary variable was created for each participant with 1 for the responder and 0 for the non nonresponder at each visit. Week 1 was considered as the Baseline. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline was set to missing as well. Change from Baseline of Week 16 and Week 24 are incorporated here which are Follow up weeks.
Time Frame: Week 16 and 24
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: mL
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
mL
  Week 16: number analyzed (Participants) | 94 | 89
  Week 16 | 0.109 (0.0345) | 0.010 (0.0392)
  Week 24: number analyzed (Participants) | 97 | 96
  Week 24 | 0.065 (0.0356) | -0.021 (0.0368)

6. Secondary Outcome: Percentage of Participants Who Demonstrated a Clinically Meaningful Increase in FEV1 Over the 12 Week Assessment Period
Description: FEV1 is forced expiratory volume in 1 second.A participant is defined as a FEV1 responder if he/she achieves a change from baseline FEV1 of >=200ml. To evaluate whether the participant was a responder over 12 weeks, change from baseline FEV1 over 12 weeks was calculated by taking the mean of the changes at Visit 7, Visit 9 and Visit 11. A binary variable was created for each participant with 1 for the responder and 0 for the non-responder. If either Visit 9 or Visit 11 FEV1 data are missing, then the binary variable for the responder over 12 weeks was set to be missing. If Visit 7 data were missing, but Visit 9 and Visit 11 data were available, then the binary variable for the responder over 12 weeks was still calculated.
Time Frame: Upto 12 weeks
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Percentage of Participants
  Week 2: number analyzed (Participants) | 98 | 97
  Week 2 | 16 | 20
  Week 4: number analyzed (Participants) | 96 | 93
  Week 4 | 22 | 23
  Week 8: number analyzed (Participants) | 93 | 91
  Week 8 | 25 | 15
  Week 12: number analyzed (Participants) | 91 | 90
  Week 12 | 34 | 20

7. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Up to Week 25
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Participants
  Any AEs | 49 | 52
  Any SAEs | 5 | 8

8. Secondary Outcome: Number of Participants With Abnormal Vital Signs of Potential Clinical Importance: Systolic and Distolic Blood Pressure and Heart Rate.
Description: Vital signs including systolic and diastolic blood pressure and heart rate taken at certain visits from screening to follow-up. Potential Clinical Importance Ranges were systolic blood pressure (<85 and >160millimeter of mercury [mmHg]), diastolic blood pressure (<45 and >100 mmHg) and heart rate (<40 and >110 beats per minute [BPM]). Number of participants with abnormal systolic blood pressure, diastolic blood pressure and heart rate values of potential clinical importance were summarized.
Time Frame: Screening, Day -28, 1, 15, 29, 50, 57 and 169 (follow-up 3)
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Participants
  Systolic Blood Pressure, High | 6 | 6
  Diastolic Blood Pressure, High | 8 | 4
  Heart Rate | 0 | 1

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormality in 12-lead Electrocardiogram (ECG)
Description: Single 12-lead ECGs were obtained at certain visits from screening to follow-up. ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and Corrected QT (QTc) intervals. Number of participants with clinically significant abnormality in 12-lead ECG readings were summarized.
Time Frame: Upto Week 25
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Participants
  Day 29, 1.5 hours: number analyzed (Participants) | 96 | 94
  Day 29, 1.5 hours | 0 | 1
  Day 29, 6 hours: number analyzed (Participants) | 96 | 94
  Day 29, 6 hours | 0 | 1
  Day 50: number analyzed (Participants) | 81 | 83
  Day 50 | 0 | 2

10. Secondary Outcome: Number of Participants With Abnormal Hematological Parameters of Potential Clinical Importance
Description: Blood samples were collected on each visit from Week 1 to Week 25 to assess the haematological parameters. White Blood Cells count, Neutrophils, Haemoglobin, Hematocrit, Count and Lymphocytes were analyzed in haematology. Number of participants with any abnormal hematological parameters of potential clinical importance are summarized here.
Time Frame: Upto Week 25
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Participants
  Low lymphocyte count | 5 | 3
  Increased white blood cell count | 3 | 1
  Low neutrophils count | 3 | 4
  Low platelet count | 1 | 1

11. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry Parameters of Potential Clinical Importance
Description: Blood samples were collected on each visit from Week 1 to Week 25 to assess the clinical chemistry parameters. Albumin, Calcium, Glucose, Pottasium, Sodium and Total Carbon Di-oxide were analyzed in clinical chemistry. Number of participants with any abnormal clinical chemistry parameters of potential clinical importance are summarized here.
Time Frame: Upto Week 25
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Participants
  Low total carbondioxide | 14 | 17
  High glucose | 10 | 17
  Low glucose | 4 | 3
  Increased total bilirubin | 2 | 2
  Increased AST | 1 | 2
  Increased ALT | 2 | 1
  Increased alkaline phosphatase | 1 | 0
  Increased serum potassium | 0 | 2
  Increased serum calcium | 1 | 0

12. Secondary Outcome: Number of Participants With Abnormal Urinanalysis Parameters of Potential Clinical Importance
Description: Samples were collected on each visit from Week 1 to Week 25 for urinalysis. Number of participants with any abnormal urinalysis parameters of potential clinical importance are summarized here.
Time Frame: Upto Week 25
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Participants | 0 | 0

13. Secondary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Concentration-time Curve Over the Dosing Interval (AUC (0-τ)).
Description: Plasma concentration-time data were well described by a 2-compartment model with first order elimination. Plasma concentrations of GSK679586 were determined at Day 1 (Pre-dose, 0.25h, 1.00h), Day 4 (72h), Day 29 (672 h), Day 57 (1344h), Day 61 (1440h), Day 85 (2016h), Day 141 (3360h), Day 169 (4032h) and Follow up visits. However, the derived PK parameters were determined only for the day of infusion administration. i.e. Day 1, Day 29 and Day 57. The AUC at Day 1 indicates AUC(0-1 h), Day 29 indicated AUC(0-672 h) and Day 57 indicated AUC(0-1344h). AUC(0-τ) for each participant was reconstructed from sparse PK sampling using Bayesian prediction obtained from a population PK model using nonlinear mixed effects methods (NONMEM, version V).
Time Frame: Day 1 (Pre-dose, 0.25h, 1.00h), Day 4 (72h), Day 29 (672h), Day 57 (1344h), Day 61 (1440h), Day 85 (2016h), Day 141 (3360h), Day 169 (4032h) and Follow up visits.
Population: PK Population comprised of participants in the ITT population for whom a pharmacokinetic samples were obtained and analyzed. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/mL
Arm/Group | GSK679586 10 mg/kg
Number analyzed (Participants) | 99
nanogram*hour/mL
  Day 1 | 64787259 (16.16)
  Day 29: number analyzed (Participants) | 94
  Day 29 | 86256087 (18.21)
  Day 57: number analyzed (Participants) | 92
  Day 57 | 93710588 (22.83)

14. Secondary Outcome: PK Parameter:Maximum Observed Concentration (Cmax)
Description: Plasma concentration-time data were well described by a 2-compartment model with first order elimination. Plasma concentrations of GSK679586 were determined at Day 1 (Pre-dose, 0.25h, 1.00h), Day 4 (72h), Day 29 (672h), Day 57 (1344h), Day 61 (1440h), Day 85 (2016h), Day 141 (3360h), Day 169 (4032h) and Follow up visits. However, Cmax were determined only for the day of infusion administration. i.e. Day 1, Day 29 and Day 57. The Cmax at Day 1 indicates Cmax(0-1 h), Day 29 indicated Cmax(0-672 h) and Day 57 indicated Cmax(0-1344 h). Cmax for each participant was reconstructed from sparse PK sampling using Bayesian prediction obtained from a population PK model using nonlinear mixed effects methods (NONMEM, version V).
Time Frame: Day 1 (Pre-dose, 0.25h, 1.00h), Day 4 (72h), Day 29 (672 h), Day 57 (1344h), Day 61 (1440h), Day 85 (2016h), Day 141 (3360h), Day 169 (4032h) and Follow up visits.
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/mL
Arm/Group | GSK679586 10 mg/kg
Number analyzed (Participants) | 99
nanogram (ng)/mL
  Day 1 | 278610.6 (33.40)
  Day 29: number analyzed (Participants) | 94
  Day 29 | 332528.4 (30.85)
  Day 57: number analyzed (Participants) | 92
  Day 57 | 355177.0 (30.31)

15. Secondary Outcome: PK Parameter: Systemic Clearance of Parent Drug
Description: Plasma concentration-time data were well described by a 2-compartment model with first order elimination. Plasma concentrations of GSK679586 were determined at Day 1 (Pre-dose, 0.25h, 1.00h), Day 4 (72h), Day 29 (672h), Day 57 (1344h), Day 61 (1440h), Day 85 (2016h), Day 141 (3360h), Day 169 (4032h) and Follow up visits. However, systemic clearance were determined only for the day of infusion administration. i.e. Day 1, Day 29 and Day 57. The systemic clearance at Day 1 indicates systemic clearance(0-1 h), Day 29 indicated systemic clearance(0-672 h) and Day 57 indicated systemic clearance(0-1344 h). Systemic clearance of parent drug for each participant was reconstructed from sparse PK sampling using Bayesian prediction obtained from a population PK model using nonlinear mixed effects methods (NONMEM, version V).
Time Frame: as for outcome 14
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/kg
Arm/Group | GSK679586 10 mg/kg
Number analyzed (Participants) | 99
L/h/kg
  Day 1 | 0.00010 (22.76)
  Day 29: number analyzed (Participants) | 94
  Day 29 | 0.00010 (22.28)
  Day 57: number analyzed (Participants) | 92
  Day 57 | 0.00010 (22.48)

16. Secondary Outcome: PK Parameter: Volume of Distribution
Description: Plasma concentration-time data were well described by a 2-compartment model with first order elimination. Plasma concentrations of GSK679586 were determined at Day 1 (Pre-dose, 0.25h, 1.00h), Day 4 (72h), Day 29 (672 h), Day 57 (1344h), Day 61 (1440h), Day 85 (2016h), Day 141 (3360h), Day 169 (4032h) and Follow up visits. However, volume of distribution were determined only for the day of infusion administration. i.e. Day 1, Day 29 and Day 57. The volume of distribution at Day 1 indicates volume of distribution(0-1 h), Day 29 indicated volume of distribution (0-672 h) and Day 57 indicated volume of distribution (0-1344 h). Volume of distribution for each participant was reconstructed from sparse PK sampling using Bayesian prediction obtained from a population PK model using nonlinear mixed effects methods (NONMEM, version V). The 2-compartment model provided the data for volume of distribution of central compartment (V1) and volume distribution of peripheral compartment (V2).
Time Frame: as for outcome 14
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/Kg
Arm/Group | GSK679586 10 mg/kg
Number analyzed (Participants) | 99
L/Kg
  V1, Day 1 | 0.0356 (33.73)
  V1, Day 29: number analyzed (Participants) | 94
  V1, Day 29 | 0.0355 (34.43)
  V1, Day 57: number analyzed (Participants) | 92
  V1, Day 57 | 0.0354 (34.77)
  V2, Day 1 | 0.0296 (0.00)
  V2, Day 29: number analyzed (Participants) | 94
  V2, Day 29 | 0.0296 (0.00)
  V2, Day 57: number analyzed (Participants) | 92
  V2, Day 57 | 0.0296 (0.00)

17. Secondary Outcome: Number of Participants With Confirmed Positive Anti-GSK679586 Antibody Results After Initiation of Study Treatment
Description: Serum samples were tested for presence of anti-GSK679586 antibodies. Blood samples were collected via an indwelling cannula or by direct venepuncture collected into a serum separator tube and allowed to clot for 1 to 2 hours. Samples were centrifuged and the resultant serum was transferred to 3 separate cryovials and stored at -80°C until shipped on dry ice to the central laboratory. Samples were analyzed in a tiered assay format. Number of participants with confirmed positive Anti-GSK679586 antibody results after initiation of study treatment were reported.
Time Frame: Up to Week 25
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK679586 10 mg/kg
Number analyzed (Participants) | 99 | 99
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: All SAEs and Non-SAE were collected from Screening (Week -8) to Follow-up Visit 3 (Week 25).
Description: SAEs were reported on ITT population
Arm/Group | Placebo | GSK679586 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/99 | 1/99
Serious Adverse Events (participants affected / at risk) | 5/99 | 8/99
Other Adverse Events (participants affected / at risk) | 19/99 | 27/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=99) | GSK679586 10 mg/kg (N=99)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cholesystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Narcotic intoxication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Rectal haemorrhage/ (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=99) | GSK679586 10 mg/kg (N=99)
Nasopharyngitis (Infections and infestations) | 5 (5) | 10 (11)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 4 (5)
Pharyngitis (Infections and infestations) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 6 (7) | 13 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.